CLINICAL TRIAL: NCT02313792
Title: Efficacy, Safety and Quality of Life of Palifermin on Reducing Oral Mucositis in Patients With Hematopoietic Stem Cell Transplantation, Prospective Double-blind Randomized Phase III Trial
Brief Title: Palifermin for Patients Receiving Hematopoietic Stem Cell Transplantation
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Catholic University of Korea (Other)
Collaborators: BLNH (Unknown)
Responsible Party: Principal Investigator, Ki-Seong Eom, MD, Associate Professor, The Catholic University of Korea
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CBMTC-supp002
Record Dates: First submitted 2014-12-05; First posted 2014-12-10 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Mucositis
Keywords: Hematopoietic stem cell transplantation; Palifermin
MeSH Terms: conditions — Mucositis | interventions — Fibroblast Growth Factor 7

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Palifermin (Active Comparator): The patients belong to this arm will be given palifermin, keratinocyte growth factor, in addition to the conventional supportive care for oral mucositis. Palifermin will be given at a dose of 60 mcg/kg for 3 days before commencement of the preparative regimen and for 3 days after stem cell infusion
  Interventions: Drug: Palifermin
- Normal saline (Placebo Comparator): The patients belong to this arm will be given normal saline as placebo plus conventional supportive care for oral mucositis. Normal saline will be given at the same volume and schedule with the study drug.

INTERVENTIONS:
Drug: Palifermin
  Arms: Palifermin

SUMMARY:
The purpose of this study is to compare the efficacy and safety of palifermin on reducing mucositis for patients receiving autologous or allogeneic stem cell transplantation with supportive care.

ELIGIBILITY:
Inclusion Criteria:

* adequate organ function
* patients who will receive autologous stem cell transplantation
* patients who will receive allogeneic stem cell transplantation using myeloablative conditioning regimen

Exclusion Criteria:

* presence of concomitant malignancy
* presence of active infection or oral mucositis prior to stem cell transplantation
* any conditions where the severity of oral mucositis cannot be evaluated

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-03 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Duration of severe oral mucositis after stem cell transplantation | 5 weeks
  from onset of severe oral mucositis till resolution of the mucositis or 28 days after stem cell transplantation

SECONDARY OUTCOMES:
Incidence of severe oral mucositis after stem cell transplantation | 5 weeks
  from onset of severe oral mucositis till resolution of the mucositis or 28 days after stem cell transplantation
Average VAS score during severe oral mucositis | 5 weeks
  from onset of severe oral mucositis till resolution of the mucositis or 28 days after stem cell transplantation
Requirement of opioid drugs during severe oral mucositis | 5 weeks
  from onset of severe oral mucositis till resolution of the mucositis or 28 days after stem cell transplantation
Requirement of opioid drugs | 5 weeks
  from onset of severe oral mucositis till resolution of the mucositis or 28 days after stem cell transplantation
Cost effectiveness of palifermin during stem cell transplantation | 5 weeks
  from admission for stem cell transplantation to discharge
Quality of life during transplant period | 5 weeks
  1 week before stem cell infusion to discharge